CLINICAL TRIAL: NCT03419403
Title: Phase 3b Study for Management of Ocular Side Effects in Subjects With EGFR-amplified Glioblastoma Receiving Depatuxizumab Mafodotin (ABT-414)
Brief Title: UNITE Study: Understanding New Interventions With GBM ThErapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated because clinical development of depatuxizumab mafodotin in glioblastoma was stopped due to lack of survival benefit.
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16-534; 2017-003171-64 (EudraCT Number)
Expanded Access: NCT03123952 (No longer available)
Record Dates: First submitted 2018-01-26; First posted 2018-02-05 (Actual); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme (GBM); Cancer; Chemoradiation therapy; Epidermal growth factor receptor-amplified glioblastoma; Radiation; Temozolomide
MeSH Terms: conditions — Glioblastoma; Neoplasms | interventions — depatuxizumab mafodotin; ABT-414; Temozolomide; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard Steroids (Experimental): Steroid eye drops: 1 drop each eye, 3 times/day, starting 2 days prior to depatuxizumab mafodotin infusion and continuing until 4 days after infusion, for a total of 7 days
  Interventions: Drug: Steroid eye drops; Drug: Depatuxizumab mafodotin; Drug: Temozolomide; Radiation: Radiation
- Standard Steroids + Vasoconstrictor + Cold Compress (Experimental): Steroid eye drops: 1 drop each eye, 3 times/day, starting 2 days prior to depatuxizumab mafodotin infusion and continuing until 4 days after infusion, for a total of 7 days; Vasoconstrictor Eye Drops: 1 drop each eye 4 - 6 times on day of infusion in total (5 - 10 minutes before infusion; at end of infusion; and 2 - 4 times during the remainder of the infusion day). Continuing 4 - 6 times/day on Day 1 and Day 2 after each depatuxizumab mafodotin infusion; Cold Compress: Starting 5 minutes prior to start of infusion and continuing for 30 minutes past end of infusion, and then use at least 2 hours total/day on Days 1 - 3 with each depatuxizumab mafodotin infusion. The cold compress was to be applied in increments no longer than 30 min (could be shorter if the participant was uncomfortable).
  Interventions: Drug: Steroid eye drops; Drug: Vasoconstrictor eye drops; Other: Cold compress; Drug: Depatuxizumab mafodotin; Drug: Temozolomide; Radiation: Radiation
- Enhanced Steroids + Vasoconstrictor + Cold Compress (Experimental): Enhanced steroid eye drops: 1 drop each eye, 6 times/day, starting 2 days prior to depatuxizumab mafodotin infusion and continuing until 4 days after infusion, for a total of 7 days; Ophthalmic Steroid Ointment; applied to each eye once daily before sleep, starting 2 days prior to depatuxizumab mafodotin infusion and continuing until 4 days after infusion, for a total of 7 days; Vasoconstrictor Eye Drops: 1 drop each eye 4 - 6 times on day of infusion in total (5 - 10 minutes before infusion; at end of infusion; and 2 - 4 times during the remainder of the infusion day). Continuing 4 - 6 times/day on Day 1 and Day 2 after each depatuxizumab mafodotin infusion; Cold Compress: Starting 5 minutes prior to start of infusion and continuing for 30 minutes past end of infusion, and then use at least 2 hours total/day on Days 1 - 3 with each depatuxizumab mafodotin infusion. Cold compress was to be applied in increments no longer than 30 min (could be shorter if the patient is uncomfortable).
  Interventions: Drug: Steroid eye drops; Drug: Vasoconstrictor eye drops; Other: Cold compress; Drug: Ophthalmic steroid ointment; Drug: Depatuxizumab mafodotin; Drug: Temozolomide; Radiation: Radiation

INTERVENTIONS:
Drug: Steroid eye drops — Solution, eye drop
Drug: Vasoconstrictor eye drops — Solution, eye drop
  Arms: Enhanced Steroids + Vasoconstrictor + Cold Compress; Standard Steroids + Vasoconstrictor + Cold Compress
Other: Cold compress — Cold compress
  Arms: Enhanced Steroids + Vasoconstrictor + Cold Compress; Standard Steroids + Vasoconstrictor + Cold Compress
Drug: Ophthalmic steroid ointment — Ointment
  Arms: Enhanced Steroids + Vasoconstrictor + Cold Compress
Drug: Depatuxizumab mafodotin — During the Chemoradiation Phase, participants were to receive depatuxizumab mafodotin at 2.0 mg/kg IV infusion over 30 - 40 minutes once every 2 weeks (Day 1 of Weeks 1, 3, and 5 of the 6-week regimen). During the Adjuvant Therapy Phase, participants were to receive depatuxizumab mafodotin at 1.25 mg/kg on Day 1 (± 2 days) and Day 15 (± 2 days) of each 28-day cycle as a 30 - 40 minute infusion for 12 cycles.
  Other Names: ABT-414
Drug: Temozolomide — Temozolomide was to be administered according to the local standard of care. Duration of treatment was to be 6 - 12 cycles in the adjuvant phase and at the discretion of the investigator as supported by local standard of care.
Radiation: Radiation — Radiation therapy treatment planning and administration was to be performed as per local institutional guidelines.

SUMMARY:
The objective of this study was to evaluate the effect of several ophthalmologic prophylactic treatment strategies for the management of ocular side effects (OSEs) in participants with epidermal growth factor receptor (EGFR)-amplified glioblastoma (GBM) who were being treated with depatuxizumab mafodotin (ABT-414).

DETAILED DESCRIPTION:
This Phase 3b open-label, randomized, exploratory study included 2 phases during the treatment period: chemoradiation therapy (radiation plus temozolomide [RT/TMZ]) and adjuvant therapy (TMZ). All participants received depatuxizumab mafodotin during both phases of the treatment period plus 1 of 3 prophylactic ophthalmologic treatments (standard steroids; standard steroids with vasoconstrictors and cold compress; and enhanced steroids with vasoconstrictors and cold compress. The study comprised a screening period of up to 7 weeks after surgery, a 6-week concomitant Chemoradiation Phase, an Adjuvant Phase beginning approximately 4 weeks after completion of chemoradiation, and a Follow-Up Phase.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed glioblastoma (GBM) histologically proven, World Health Organization (WHO) grade IV GBM or WHO grade IV gliosarcoma
* Tumors must demonstrate epidermal growth factor receptor (EGFR) amplification
* Tumors must be supratentorial in location
* Participant must have recovered from the effects of surgery, postoperative infection, and other complications; has no significant post-operative hemorrhage
* Participant has a Karnofsky performance status (KPS) of 70 or higher
* Participant has adequate bone marrow, renal, and hepatic function
* Electrocardiogram without evidence of acute cardiac ischemia ≤ 21 days prior to randomization
* Participant has a life expectancy of ≥ 3 months

Exclusion Criteria:

* Participant has received prior chemotherapy or radiotherapy for cancer of the head and neck region
* Participant has received prior treatment with Gliadel wafers or any other intratumoral or intracavitary treatment
* Participant has hypersensitivity to any component of temozolomide or dacarbazine
* Participant has received anti-cancer therapy (including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic, or any investigational therapy) within 5 years of Study Day 1
* Participant has clinically significant uncontrolled condition(s) as described in the protocol
* Participant has any medical condition which in the opinion of the investigator places the participant at an unacceptably high risk for toxicities
* Participant has had another active malignancy within the past 3 years except for any cancer considered cured or non-melanoma carcinoma of the skin
* Participant has a history of herpetic keratitis
* Participant is not suitable for receiving ocular steroids with conditions as described in the protocol
* Participant has had laser-assisted in situ keratomileusis (LASIK) procedure within the last 1 year or cataract surgery within the last 3 months
* Participant has a visual condition that compromises the ability to accurately measure visual acuity or assess visual activities of daily living (vADLs)
* Participant has hepatitis B virus or hepatitis C virus infection
* Participant not receiving treatment with highly active antiretroviral therapy (HAART) when positive for human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (22):
- United States (9):
  - Usc /Id# 164235, Los Angeles, California
  - Moffitt Cancer Center /ID# 164234, Tampa, Florida
  - Rush University Medical Center /ID# 171003, Chicago, Illinois
  - Northshore University Health System-Evanston /ID# 164221, Evanston, Illinois
  - CDH-Delnor Health System /ID# 169909, Warrenville, Illinois
  - Columbia University Medical Center /ID# 164220, New York, New York
  - Levine Cancer Ins, Carolina Me /ID# 171271, Charlotte, North Carolina
  - UT Health Science Ctr-Houston /ID# 164223, Houston, Texas
  - Baylor Scott & White Medical Center- Temple /ID# 170792, Temple, Texas
- Australia (4):
  - Royal North Shore Hospital /ID# 169673, Saint Leonards, New South Wales
  - Calvary Mater Newcastle /ID# 169672, Waratah, New South Wales
  - Royal Brisbane and Women's Hospital /ID# 169674, Herston, Queensland
  - Austin Hospital /ID# 169671, Heidelberg, Victoria
- Germany (4):
  - Universitaetsklinik Heidelberg /ID# 169970, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Leipzig /ID# 169969, Leipzig, Saxony
  - Klinikum Univ. Regensburg /ID# 169963, Regensburg
  - Universitatsklinikum Tubingen /ID# 169965, Tübingen
- Netherlands (2):
  - Vrije Universiteit Medisch Centrum /ID# 170152, Amsterdam
  - Universitair Medisch Centrum Utrecht /ID# 170149, Utrecht
- United Kingdom (3):
  - Guy's and St Thomas' NHS Found /ID# 207752, London, London, City of
  - Queen Elizabeth Hospital - BIRMINGHAM /ID# 200657, Birmingham
  - Castle Hill Hospital /ID# 200662, Cottingham

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All randomized participants
Groups:
- Untreated Participants: Participants who were randomized to the study but received no doses of depatuxizumab mafodotin or prophylactic eye treatments
Period: Overall Study
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress | Untreated Participants
Started | 14 | 12 | 12 | 2
Completed | 2 | 3 | 0 | 0
Not Completed | 12 | 9 | 12 | 2
Not completed — Withdrawal by Subject | 5 | 2 | 5 | 1
Not completed — Progressive disease (per protocol) | 0 | 2 | 2 | 0
Not completed — Other, not specified | 6 | 4 | 5 | 1
Not completed — Left study due to COVID-19 restrictions | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: All randomized participants who received at least 1 dose of depatuxizumab mafodotin
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress | Total
Number analyzed (Participants) | 14 | 12 | 12 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.85) | 55.2 (10.53) | 57.3 (8.69) | 53.1 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 8
  Male | 11 | 8 | 11 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 12 | 12 | 36
  Black or African American | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Required a Change in Ocular Side Effect (OSE) Management
Description: Inadequate control of ocular side effects (OSE) was defined as either a ≥ 3-line decline from baseline (≥ +0.3 on LogMAR scale) in visual acuity (with baseline correction determined at the screening ophthalmology visit)) or ≥ Grade 3 OSE severity on the Corneal Epithelial Adverse Event (CEAE) scale.
Time Frame: Within 8 weeks after the initial dose of depatuxizumab mafodotin
Population: Safety population: all randomized participants who received at least 1 dose of depatuxizumab mafodotin and had at least 1 post-baseline assessment within 8 weeks after the initial dose for either LogMAR or CEAE
Measure: Number; unit: percentage of participants
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 14 | 12 | 12
percentage of participants
  Bilateral vision | 50.0 | 27.3 | 41.7
  Vision in worst eye | 64.3 | 72.7 | 50.0

2. Secondary Outcome: Maximum Change From Baseline on the Logarithm of the Minimum Angle of Resolution (LogMAR) Scale
Description: The LogMAR scale measures visual acuity on a continuous scale, with a LogMAR value of 0 equivalent to 20/20 visual acuity. Normal vision is considered to be from -0.2 - 0.1; higher values indicate visual impairment. The baseline observation is defined as the last non-missing measurement collected prior to the first dose of depatuxizumab mafodotin.
Time Frame: Within 8 weeks after the initial dose of depatuxizumab mafodotin
Population: Safety population: all randomized participants who received at least 1 dose of depatuxizumab mafodotin and had available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 12 | 10 | 9
units on a scale
  Bilateral vision | 0.353 (0.1888) | 0.402 (0.1985) | 0.272 (0.3888)
  Vision in worst eye | 0.482 (0.2028) | 0.528 (0.3073) | 0.430 (0.5120)

3. Secondary Outcome: Time to Bandage Contact Lens (BCL) Intervention
Description: The time to initiation of bandage contact lenses for those participants who required intervention due to inadequate control of ocular side effects (OSE) was calculated.
Time Frame: Up to 9 months after the first dose of depatuxizumab mafodotin
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 14 | 12 | 12
months | NA [1.1 to NA] — Not calculable due to insufficient number of participants with events | 3.6 [1.1 to NA] — Not calculable due to insufficient number of participants with events | 2.1 [1.1 to NA] — Not calculable due to insufficient number of participants with events

4. Secondary Outcome: Number of Participants With Depatuxizumab Mafodotin Dose Modifications Due to Ocular Side Effects (OSE)
Description: Dose modifications included depatuxizumab mafodotin withdrawal, interruption, and reductions in dose initiated due to OSEs.
Time Frame: From the first dose of study drug until 49 days after last depatuxizumab mafodotin administration, up to 47 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 14 | 12 | 12
Participants | 2 | 3 | 2

5. Secondary Outcome: Cumulative Dose of Depatuxizumab Mafodotin Received During Chemoradiation and During Adjuvant Treatment
Description: The cumulative dose of depatuxizumab mafodotin administered was tabulated.
Time Frame: Up to 9 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 14 | 12 | 12
mg/kg | 8.5 (5.86) | 10.5 (7.35) | 7.0 (3.67)

6. Secondary Outcome: Treatment-Emergent Corneal Epithelial Adverse Event (CEAE) Grade at Each Visit
Description: The corneal epithelial adverse event (CEAE) rating scale is designed to record symptoms associated with corneal epitheliopathy caused by antibody-drug conjugates and to grade the severity of findings. The overall CEAE grade is measured on a scale of 0 to 5, with higher values being more severe, reflecting the impact of corneal abnormalities on visual activities of daily living (ADLs). Additional detailed information is collected for specific domains that are commonly affected, with the following ranges (each in order of increasing severity): ocular discomfort (0 - 4), photophobia (0 - 3), and reading (1 - 3).
Time Frame: Up to 47 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 14 | 12 | 12
Participants
  Week 1: Grade 0 | 10 | 8 | 5
  Week 1: Grade 1 | 1 | 3 | 1
  Week 3: Grade 0 | 4 | 5 | 7
  Week 3: Grade 1 | 10 | 6 | 3
  Week 3: Grade 2 | 0 | 0 | 1
  Week 5: Grade 0 | 1 | 0 | 2
  Week 5: Grade 1 | 7 | 5 | 6
  Week 5: Grade 2 | 1 | 3 | 2
  Week 5: Grade 3 | 4 | 2 | 2
  Week 7: Grade 0 | 0 | 0 | 2
  Week 7: Grade 1 | 3 | 4 | 0
  Week 7: Grade 2 | 4 | 6 | 5
  Week 7: Grade 3 | 2 | 0 | 2
  Week 9: Grade 0 | 1 | 0 | 1
  Week 9: Grade 1 | 1 | 2 | 0
  Week 9: Grade 2 | 3 | 5 | 4
  Week 9: Grade 3 | 2 | 0 | 1
  Week 11: Grade 0 | 0 | 0 | 1
  Week 11: Grade 1 | 2 | 1 | 0
  Week 11: Grade 2 | 2 | 0 | 3
  Week 11: Grade 3 | 1 | 0 | 1
  Week 11: Grade 4 | 1 | 0 | 0
  Week 13: Grade 1 | 1 | 0 | 1
  Adj Week 1: Grade 0 | 0 | 1 | 0
  Adj Week 1: Grade 1 | 1 | 3 | 2
  Adj Week 1: Grade 2 | 3 | 2 | 2
  Adj Week 1: Grade 3 | 1 | 0 | 0
  Adj Week 5: Grade 0 | 0 | 2 | 2
  Adj Week 5: Grade 1 | 1 | 3 | 0
  Adj Week 5: Grade 2 | 4 | 0 | 1
  Adj Week 5: Grade 3 | 1 | 1 | 0
  Adj Week 9: Grade 0 | 0 | 1 | 0
  Adj Week 9: Grade 1 | 0 | 2 | 1
  Adj Week 9: Grade 2 | 2 | 2 | 2
  Adj Week 9: Grade 3 | 1 | 1 | 0
  Adj Week 13: Grade 0 | 0 | 1 | 0
  Adj Week 13: Grade 1 | 0 | 2 | 0
  Adj Week 13: Grade 2 | 2 | 2 | 2
  Adj Week 13: Grade 3 | 1 | 0 | 0
  Adj Week 17: Grade 0 | 0 | 0 | 1
  Adj Week 17: Grade 1 | 0 | 1 | 0
  Adj Week 17: Grade 2 | 2 | 3 | 0
  Adj Week 21: Grade 1 | 0 | 0 | 1
  Adj Week 21: Grade 2 | 2 | 3 | 0
  Adj Week 25: Grade 1 | 0 | 2 | 0
  Adj Week 25: Grade 2 | 1 | 1 | 0
  Adj Week 29: Grade 2 | 1 | 0 | 0
  Adj Week 29: Grade 4 | 0 | 1 | 0

7. Secondary Outcome: Change From Baseline In Logarithm of the Minimum Angle of Resolution (LogMAR) Scale After Bandage Contact Lens (BCL) Intervention
Description: The change on the LogMAR Scale from last assessment prior to BCL intervention to 2 weeks after BCL intervention was calculated. The LogMAR scale measures visual acuity on a continuous scale, with a LogMAR value of 0 equivalent to 20/20 visual acuity. Normal vision is considered to be from -0.2 - 0.1; higher values indicate visual impairment.
Time Frame: From the last assessment prior to BCL intervention to 2 weeks after BCL intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 4 | 2 | 3
units on a scale
  Within 8 weeks of first dose: Bilateral vision | 0.325 (0.1248) | 0.13 (0.099) | 0.54 (0.1442)
  Within 8 weeks of first dose: Vision in worst eye | 0.435 (0.0574) | 0.52 (0.3111) | 0.867 (0.2914)
  Within 8 weeks of first adjuvant dose: Bilateral vision: number analyzed (Participants) | 1 | 2 | 0
  Within 8 weeks of first adjuvant dose: Bilateral vision | -0.1 | 0.41 (0.2404) |
  Within 8 weeks of first adjuvant dose: Vision in worst eye: number analyzed (Participants) | 1 | 2 | 0
  Within 8 weeks of first adjuvant dose: Vision in worst eye | -0.1 | 0.33 (0.0141) |

8. Secondary Outcome: Percentage of Participants That Recovered to <3-line Decline From Baseline (≤ +0.3 LogMAR) in Visual Acuity After Bandage Contact Lens (BCL) Intervention
Description: Recovery was defined as return to <3-line decline from baseline (≤ +0.3 LogMAR) in visual acuity after BCL intervention.
Time Frame: From the last assessment prior to BCL intervention to the end of BCL intervention
Population: Data were not collected for this outcome (due to early termination of the study).
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Depatuxizumab Mafodotin Dose Modifications to Ocular Side Effects After Bandage Contact Lens (BCL) Intervention
Description: Dose modifications included depatuxizumab mafodotin withdrawal, interruption, and reductions in dose initiated due to OSEs after BCL intervention.
Time Frame: From the last assessment prior to BCL intervention to the end of BCL intervention, up to 38 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 14 | 12 | 12
participants | 2 | 1 | 0

10. Secondary Outcome: Time to Restart Depatuxizumab Mafodotin if Interrupted Due to Ocular Side Effects After Bandage Contact Lens (BCL) Intervention
Description: The time to restart depatuxizumab mafodotin treatment if it was interrupted due to ocular side effects after BCL Intervention was tabulated.
Time Frame: From the last assessment prior to BCL intervention to the end of BCL intervention
Population: Data were not collected for this outcome (due to early termination of the study).
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Treatment Emergent Corneal Epithelial Adverse Event (CEAE) Grade at Each Visit After Bandage Contact Lens (BCL) Intervention
Description: as for outcome 6
Time Frame: From the last assessment prior to BCL intervention to the end of BCL intervention, up to 38 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 7 | 4 | 4
Participants
  Week 5: Grade 1 | 2 | 0 | 0
  Week 7: Grade 2 | 1 | 1 | 0
  Week 9: Grade 2 | 1 | 1 | 1
  Week 11: Grade 2 | 0 | 0 | 2
  Week 11: Grade 3 | 1 | 0 | 0
  Week 13: Grade 1 | 1 | 0 | 0
  Adj Week 1: Grade 1 | 0 | 0 | 1
  Adj Week 1: Grade 2 | 0 | 0 | 1
  Adj Week 5: Grade 0 | 0 | 1 | 1
  Adj Week 5: Grade 1 | 0 | 1 | 0
  Adj Week 5: Grade 2 | 1 | 0 | 1
  Adj Week 5: Grade 3 | 1 | 0 | 0
  Adj Week 9: Grade 0 | 0 | 1 | 0
  Adj Week 9: Grade 1 | 0 | 0 | 1
  Adj Week 9: Grade 2 | 0 | 0 | 1
  Adj Week 9: Grade 3 | 1 | 0 | 0
  Adj Week 13: Grade 0 | 0 | 2 | 0
  Adj Week 13: Grade 1 | 0 | 1 | 0
  Adj Week 13: Grade 2 | 1 | 0 | 1
  Adj Week 13: Grade 3 | 1 | 0 | 0
  Adj Week 17: Grade 1 | 0 | 1 | 0
  Adj Week 17: Grade 2 | 1 | 1 | 0
  Adj Week 21: Grade 2 | 2 | 1 | 0
  Adj Week 25: Grade 1 | 0 | 1 | 0
  Adj Week 25: Grade 2 | 1 | 0 | 0
  Adj Week 29: Grade 2 | 1 | 0 | 0

12. Secondary Outcome: Time to Ocular Side Effect (OSE) Symptom Resolution After Drug Discontinuation (Reversibility)
Description: The time from discontinuation of depatuxizumab mafodotin to OSE symptom resolution (reversibility) was to be recorded.
Time Frame: From the first dose of study drug until 49 days after last depatuxizumab mafodotin administration, up to 47 weeks
Population: Data were not collected for this outcome (due to early termination of the study).
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Time to Re-initiation of Depatuxizumab Mafodotin After Dose Interruption
Description: The time from dose interruption until re-initiation or permanent discontinuation of depatuxizumab mafodotin was to be recorded.
Time Frame: Up to 9 months
Population: Data were not collected for this outcome (due to early termination of the study).
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 49 days after last depatuxizumab mafodotin administration, up to 47 weeks. In addition, serious adverse events and protocol-related nonserious adverse events were collected from the time the participant signed the study-specific informed consent.
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time that the first dose of depatuxizumab mafodotin is administered until 49 days have elapsed following discontinuation of study drug. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Standard Steroids | Standard Steroids + Vasoconstrictor + Cold Compress | Enhanced Steroids + Vasoconstrictor + Cold Compress
All-Cause Mortality (participants affected / at risk) | 1/14 | 1/12 | 1/12
Serious Adverse Events (participants affected / at risk) | 6/14 | 4/12 | 4/12
Other Adverse Events (participants affected / at risk) | 14/14 | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Steroids (N=14) | Standard Steroids + Vasoconstrictor + Cold Compress (N=12) | Enhanced Steroids + Vasoconstrictor + Cold Compress (N=12)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
ULCERATIVE KERATITIS (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
EYE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
TUMOUR PSEUDOPROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
STATUS EPILEPTICUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Steroids (N=14) | Standard Steroids + Vasoconstrictor + Cold Compress (N=12) | Enhanced Steroids + Vasoconstrictor + Cold Compress (N=12)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 1 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (4) | 5 (7) | 3 (7)
CARDIOMEGALY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0)
ACQUIRED EPIBLEPHARON (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
DIPLOPIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
EYELID PTOSIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
FOREIGN BODY SENSATION IN EYES (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 5 (5) | 4 (4) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 6 (7) | 6 (7) | 3 (3)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 6 (10) | 9 (10) | 7 (8)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (2) | 0 (0) | 0 (0)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 2 (3) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
BALANITIS CANDIDA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (1)
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
RADIATION NECROSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 5 (7) | 3 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4) | 2 (2) | 2 (3)
BLOOD BILIRUBIN ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD CALCIUM INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
CARDIAC MURMUR (Investigations) | 0 (0) | 0 (0) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 3 (7)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
NEUTROPHIL COUNT INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (2) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (2) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 (4) | 3 (5) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
APRAXIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (3) | 1 (1)
HEADACHE (Nervous system disorders) | 5 (5) | 3 (3) | 4 (5)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3)
SYNCOPE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
VASOGENIC CEREBRAL OEDEMA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
ANXIETY (Psychiatric disorders) | 0 (0) | 2 (3) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 5 (7)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SCAR PAIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT03419403/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03419403/SAP_001.pdf